CLINICAL TRIAL: NCT02483572
Title: Treatment of Severe Destructive Behavior: Functional Communication Training Versus Wait-List Control
Brief Title: Treatment of Severe Destructive Behavior: FCT Versus Wait-List Control
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to maintain a waitlist long enough to serve as a control group.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0363-15-FB
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Aggression; Self-Injurious Behavior
MeSH Terms: conditions — Aggression; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Communication Training (Experimental): Participants assigned to this condition will receive treatment immediately after assignment. The investigators will implement functional communication training (FCT) to teach the participant an appropriate request response, known as a functional communication response or FCR. FCT training will continue until the participant emits independent FCRs in at least 90% of the 30-s intervals and until destructive behavior decreases by 90% (relative to pre-treatment baseline) for two consecutive sessions.
  Interventions: Behavioral: Functional Communication Training
- Waitlist-Control Condition (No Intervention): Participants assigned to the waitlist-control condition will not immediately receive services. These participants will be paired with an FCT-condition participant such that the no-treatment duration for these participants is yoked to the amount of time their respective FCT-condition participants receive services (e.g., most treatment last approximately 4 months, or 16 weeks); if Participant A finishes treatment in 16 weeks, Participant B will not receive treatment for at least 16 weeks for comparative measures). After the wait period, these participants will then receive the same services as those assigned to the immediate treatment (FCT Condition).

INTERVENTIONS:
Behavioral: Functional Communication Training — Functional communication training (FCT) is the most widely used treatment for severe destructive behavior that is maintained by social reinforcement, such as access to attention, tangible items, or escape from nonpreferred activities. Once clinicians determine the functional reinforcer for destructive behavior, the clinician can then teach the child an appropriate, functionally-equivalent response (e.g., exchanging a card to access parental attention) and the clinician would no longer provide the functional reinforcer for destructive behavior.
  Arms: Functional Communication Training

SUMMARY:
Children with an intellectual disability often display severe destructive behavior (e.g., aggression, self-injury) that pose risks to themselves or others and represent barriers to community integration. Destructive behaviors are often treated with behavioral interventions derived from a functional analysis, which is used to identify the antecedents and consequences that occasion and reinforce the destructive behavior. One treatment is called functional communication training (FCT), which involves extinction of destructive behavior and reinforcement of an alternative communication response with the consequence that previously reinforced destructive behavior. Results from epidemiological studies and meta-analyses indicate that treatments based on functional analysis, like FCT, typically reduce destructive behavior by 90% or more and are more effective than other treatments. However, many if not all of these studies have used within-subject experimental designs to demonstrate control of the treatment effects. Replication of the effects of FCT is typically shown on a subject-by-subject basis with relatively small numbers of patients (e.g., one to four patients). No study has demonstrated the effectiveness of FCT for treatment of destructive behavior across a large group of children.

The goal of this study is to compare FCT (which is used clinically with the majority of the investigators' patients and is considered best practice for treating destructive behavior that occurs for social reasons [e.g., to access attention, preferred toys, or to escape from unpleasant activities]) to a waitlist control group across a large number of children with destructive behavior to evaluate the generality of FCT effectiveness. The investigators will evaluate rates of destructive behavior with each patient during a pretest baseline and again following FCT (approximately four months later) and/or the waitlist control duration (again, approximately four months later). All children assigned to the waitlist-control condition will be offered FCT services by the investigators' clinic at the end of the four-month waitlist period. These children will again be tested following four months of FCT (i.e., posttest). Therefore, children assigned to the FCT condition will be tested twice (one pretest and one posttest), and children assigned to the waitlist-control condition will be tested thrice (one pretest, a second pretest following a four-month waitlist period, and one posttest).

DETAILED DESCRIPTION:
The purpose of the current investigation is to evaluate the generality of FCT as treatment for severe destructive behavior. Again, the effectiveness of FCT in treating destructive behavior has been demonstrated repeatedly both in the investigators' clinic and in other clinics. The investigators are specifically interested in examining the percentage of this population that might benefit from FCT, as well as identifying the subject characteristics of children for whom FCT is and is not effective.

Children with an intellectual disability often display severe destructive behaviors (e.g., aggression, self-injury) that pose significant risks to self or others and represent overwhelming barriers to community integration. These destructive behaviors are often treated with behavioral interventions derived from a functional analysis, which is used to identify the environmental antecedents and consequences that occasion and reinforce the destructive behavior. One such treatment is called functional communication training (FCT), which involves extinction of destructive behavior and reinforcement of an alternative communication response with the consequence that previously reinforced destructive behavior. Results from epidemiological studies and meta-analyses indicate that treatments based on functional analysis, like FCT, typically reduce destructive behavior by 90% or more and are much more effective than other treatments. Despite these impressive findings, there have been no randomized, controlled trials evaluating the effectiveness of FCT. The goal of this study is to determine the robustness of FCT in reducing severe destructive behavior as compared to a waitlist control group.

ELIGIBILITY:
Inclusion Criteria:

Child Subjects:

* Boys and girls between the ages of 3 and 18;
* Destructive behavior (e.g., aggression, property destruction, SIB) that has been the focus of outpatient behavioral and pharmacological treatment but continues to occur, on average, more than once per hour;
* Destructive behavior reinforced by social consequences (i.e., significantly higher and stable rates of the behavior in one or more social test conditions of a functional analysis [e.g., attention, escape] relative to the control condition [play] and the test condition for automatic reinforcement [alone or ignore]);
* On a stable psychoactive drug regimen (or drug free) for at least 3 months with no anticipated changes;
* Stable educational plan and placement, with no anticipated changes during the study.
* Currently enrolled or on the waiting list for the Severe Behavior Clinic.

Adult Subjects (Caregivers):

* Men and women between the ages of 19 and 70;
* Who do not have any physical limitations that would prohibit them from conducting sessions with their child (i.e., pregnant);
* Have a child who is currently enrolled or on the waiting list for the Severe Behavior Clinic.

Exclusion Criteria:

Child Subjects:

* Children not meeting the inclusion criteria above;
* Children currently receiving intensive (15 or more hours per week), function-based, behavioral treatment for their destructive behavior through the school or another program; DSM-V diagnosis of Rett syndrome or other degenerative conditions (e.g., inborn error of metabolism);
* Presence of a comorbid health condition (e.g., blindness) or major mental disorder (e.g., bipolar disorder) that would interfere with participation in the study (e.g., requiring frequent hospitalizations);
* Children with self injury who, based on the results of the risk assessment, cannot be exposed to baseline conditions without placing them at risk of serious or permanent harm (e.g., detached retinas);
* Children requiring changes in drug treatment (but such children will be invited to participate if they meet the above criteria 3 months after a stable drug regimen is achieved).

Adult Subjects (Caregivers):

* Adults who are outside the age range of 19 to 70
* Pregnant mothers (for safety purposes)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Fisher, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to make data available to participants if requested and submit results for publication
Supporting Information: Study Protocol, ICF
Time Frame: The informed consent form shall be available to the caregiver immediately after caregiver signature. If requested, the study protocol will be sent to the caregiver after the study is complete.
Access Criteria: Any caregiver enrolled in the study will be eligible to receive the above documents.

REFERENCES:
- [Background] Carr EG, Durand VM. Reducing behavior problems through functional communication training. J Appl Behav Anal. 1985 Summer;18(2):111-26. doi: 10.1901/jaba.1985.18-111. PMID 2410400
- [Background] Treatment of destructive behaviors in persons with developmental disabilities. Natl Inst Health Consens Dev Conf Consens Statement. 1989 Sep 11-13;7(9):1-14. No abstract available. PMID 2483746
- [Background] Tiger JH, Hanley GP, Bruzek J. Functional communication training: a review and practical guide. Behav Anal Pract. 2008 Spring;1(1):16-23. doi: 10.1007/BF03391716. PMID 22477675

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional Communication Training: Participants assigned to this condition will receive treatment immediately after assignment. The investigators will implement functional communication training (FCT) to teach the participant an appropriate request response, known as a functional communication response or FCR. FCT training will continue until the participant emits independent FCRs in at least 90% of the 30-s intervals and until destructive behavior decreases by 90% (relative to pre-treatment baseline) for two consecutive sessions.
  Functional Communication Training: Functional communication training (FCT) is the most widely used treatment for severe destructive behavior that is maintained by social reinforcement, such as access to attention, tangible items, or escape from nonpreferred activities. Once clinicians determine the functional reinforcer for destructive behavior, the clinician can then teach the child an appropriate, functionally-equivalent response (e.g., exchanging a card to access parental attention)
Period: Overall Study
Arm/Group | Functional Communication Training | Waitlist-Control Condition
Started | 2 | 2
Completed | 0 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Communication Training | Waitlist-Control Condition | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 6 [4 to 9] | 7 [6 to 8] | 7 [4 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Destructive behavior per min [Mean (Full Range); unit: responses per min] | 1 [.8 to 1.2] | .9 [.4 to 1.3] | .9 [.4 to 1.3]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Destructive Behavior After Treatment or Initial Wait Period
Description: The investigators will measure the rate of destructive behavior following successful treatment when implemented by participants' caregivers. Participants assigned to the wait-list control group will have their rate of destructive behavior assessed at the end of the wait period, prior to implementing treatment, to detect any changes in rate of destructive behavior due to the passage of time.
Time Frame: After treatment or initial wait period (approximately 16 weeks)
Population: We did not collect these posttest data because subjects were withdrawn prior to the posttest period (e.g., due to relocation).
Measure: Mean (Full Range); unit: responses per min
Arm/Group | Functional Communication Training | Waitlist-Control Condition
Number analyzed (Participants) | 0 | 1
responses per min |  | 2 [0 to 4.6]

2. Secondary Outcome: Rate of Functional Communication Responses (FCRs) After Treatment or Wait Period
Description: The investigators will measure the rate of functional communication responses (FCRs) following successful treatment when implemented by participants' caregivers. Participants assigned to the wait-list control group will have their rate of FCRs assessed at the end of the wait period, prior to implementing treatment, to detect any changes in rate of FCRs due to the passage of time.
Time Frame: After treatment or initial wait period (approximately 16 weeks)
Population: We withdrew both participants assigned to FCT. We completed the study with only one child assigned to the waitlist-control condition.
Measure: Mean (Full Range); unit: responses per min
Arm/Group | Functional Communication Training | Waitlist-Control Condition
Number analyzed (Participants) | 0 | 1
responses per min |  | 0 [0 to 0]

3. Secondary Outcome: Rate of Functional Communication Responses After Treatment, Following Longer Wait Period (Wait-list Control Group Only)
Description: After measuring the control group participant's rate of functional communication responses after approximately 4 months, the investigators will implement FCT treatment and assess the rate of functional communication responses following the control group participant's successful treatment (approximately 32 weeks following initial baseline). These outcome measures may demonstrate that functional communication responses exhibited by the wait-list control participants only increase to clinically significant levels following FCT treatment, rather than the passage of time.
Time Frame: End of treatment, following wait period (approximately 32 weeks)
Population: We completed the study with one child assigned to the waitlist-control condition.
Measure: Mean (Full Range); unit: responses per minute
Arm/Group | Functional Communication Training | Waitlist-Control Condition
Number analyzed (Participants) | 0 | 1
responses per minute |  | 1 [1 to 1]

4. Secondary Outcome: Rate of Destructive Behavior After Treatment, Following Longer Wait Period (Wait-list Control Group Only)
Description: After measuring the control group participant's rate of destructive behavior after approximately 4 months, the investigators will implement FCT treatment and assess the rate of destructive behavior following the control group participant's successful treatment (approximately 32 weeks following initial baseline). These outcome measures may demonstrate that destructive behavior exhibited by the wait-list control participants only reduces to clinically significant levels following FCT treatment, rather than the passage of time.
Time Frame: End of treatment, following wait period (approximately 32 weeks)
Population: Only one participant in the waitlist-control condition completed the study. We analyzed the caregiver-implemented treatment sessions for the child who completed the study.
Measure: Mean (Full Range); unit: responses per minute
Arm/Group | Functional Communication Training | Waitlist-Control Condition
Number analyzed (Participants) | 0 | 1
responses per minute |  | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: We collected data on potential adverse events over the last 3 years and 7 months.
Arm/Group | Functional Communication Training | Waitlist-Control Condition
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
We experienced two primary challenges: (1) withdrawals, both voluntary due to relocation and experimenter-led due to repeated absences and (2) too short of a waitlist to allow for pairing of subjects for a waitlist control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT02483572/Prot_SAP_000.pdf